CLINICAL TRIAL: NCT01555931
Title: Immediate vs. 4-8 Week Postpartum Levonorgestrel-releasing Intrauterine System Placement: A Randomized Clinical Trial (Short Title: PPIUD1)
Brief Title: Postpartum Levonorgestrel-releasing Intrauterine System and Breastfeeding
Acronym: PPIUD1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-1786
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2013-06

CONDITIONS: Postpartum Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate (Experimental): Placement within 48 hours of delivery
  Interventions: Drug: Levonorgestrel-releasing intrauterine system
- Control (Active Comparator): Placement 4-8 weeks after delivery
  Interventions: Drug: Levonorgestrel-releasing intrauterine system

INTERVENTIONS:
Drug: Levonorgestrel-releasing intrauterine system — Placement within 48 hours of delivery
  Other Names: Mirena

SUMMARY:
This will be a randomized clinical trial of 190 women aged 18-45 who plan to breastfeed their infant for at least 6 months and desire to use the LNG-IUS as their primary contraceptive method postpartum. The investigators will compare the frequency of breastfeeding among women receiving the levonorgestrel-releasing intrauterine system (LNG-IUS) immediately after vaginal delivery compared to 4-8 weeks later. The investigators hypothesize there will be no difference in breastfeeding prevalence between the two groups.

ELIGIBILITY:
1. Women ages 18-45
2. Pregnant and equal to or more than 24 weeks of estimated gestational age
3. States an intent to breastfeed for at least 6 months
4. States a plan to use the LNG-IUS postpartum
5. Anticipates a vaginal delivery
6. HIV negative
7. Intend to stay in the Chapel Hill area for at least 6 months after birth
8. No medical or personal conditions which in the judgment of study staff preclude participation in the study
9. Have no allergies to any component of the LNG-IUS
10. No known uterine anomalies
11. Fluent in English
12. No history of ectopic pregnancy
13. No known or suspected carcinoma of the breast
14. No known acute liver disease or liver tumor (benign or malignant)
15. No known or suspected uterine or cervical neoplasia or unresolved abnormal pap smear
16. No active pelvic inflammatory disease
17. No known hypersensitivity to any component of the LNG-IUS
18. No genital bleeding of unknown etiology
19. No history of solid organ transplantation

Additional eligibility criteria for entry into the randomized trial, as assessed postpartum

1. No endometritis or chorioamnionitis
2. Membranes ruptured for less than 24 hours prior to delivery (O'Hanley, Hayes)
3. No fever greater than or equal to 38°C during the intrapartum or postpartum period
4. Did not receive medications other than pitocin and/or misoprostol to control postpartum bleeding
5. Did not have a documented estimated blood loss of greater than 750mL intrapartum
6. Did not receive a blood transfusion for a diagnosis of postpartum hemorrhage
7. Did not have a third or fourth degree laceration at delivery.
8. The infant must be greater than 35 weeks EGA at birth as determined by physical exam at birth
9. The infant must weigh at least 2727 grams
10. Must have been a singleton birth
11. Infant not in the intensive care nursery
12. The infant has not been diagnosed with a condition which would preclude long term feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Stuart, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Women's Hospital, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 women failed entry criteria after delivery. Therefore although 61 were enrolled in the original study cohort, only 35 were randomized and allocated to one of the two treatment arms.
Period: Overall Study
Arm/Group | Immediate | Control
Started | 17 | 18
Completed | 15 | 13
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of women allocated to immediate or late LNG-IUS placement after delivery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate | Control | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25 to 30] | 27 [25 to 29] | 27 [25 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 8 | 10 | 18
  Black, non-Hispanic | 5 | 2 | 7
  Hispanic or Latina | 3 | 5 | 8
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding
Description: Reported any breastfeeding at the final 6 month visit
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Immediate | Control
Number analyzed (Participants) | 17 | 18
participants | 10 | 9

2. Secondary Outcome: LNG-IUS Expulsion or Removal
Description: Expulsion or indicated removal of the originally placed LNG-IUS at any point during the study
Time Frame: up to 6 months
Measure: Number; unit: participants
Arm/Group | Immediate | Control
Number analyzed (Participants) | 17 | 18
participants | 8 | 0

ADVERSE EVENTS:
Arm/Group | Immediate | Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No